CLINICAL TRIAL: NCT06176638
Title: Resettled Refugee Families for Healing (RRF4H): A Study of Intergenerational Impact of War Trauma and Resilience
Brief Title: Resettled Refugee Families for Healing
Acronym: RRF4H
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Nhial Timothy Tutlam, PhD, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202307081; 1K01MH131872-01A1 (NIH)
Record Dates: First submitted 2023-11-01; First posted 2023-12-20 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Stress Disorders, Post-Traumatic; Depression; Antisocial Personality Disorder; Anxiety; Aggressive Behavior
Keywords: Resettled Refugee Youth; Intergenerational Transmission of Trauma; Multiple Family Groups; TeenAge Health Consultants; Trauma-Associated Mental Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Antisocial Personality Disorder; Anxiety Disorders; Aggression

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two treatment conditions at the community level: 1) Usual Care; (2) Combination intervention consisting of: MFG + Virtual TAHC peer mentoring program. Community will be defined as geographically designated areas of Omaha, and the City of Lincoln, Nebraska. Youth in will receive the usual mental health counseling provided through their school counselors. Those in the combination intervention will receive 16 MFG sessions along with their biological parents and 16 virtual TAHC sessions with their peers (excluding parents).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RRF4H Combination Intervention Group (Experimental): This is a combination intervention that builds on the Usual Care and will consist of (1) a MFG-based FS model, which targets issues such as communication, relationship, and social support network development to assist with parenting and stress management, and stigma reduction96 and (2) a peer-mentoring program called TeenAge Health Consultants (Virtual TAHC) adapted for delivery in virtual environment.
  Interventions: Behavioral: RRF4H Combination Intervention
- Usual Care Group (No Intervention): Youth in RRF4H study will receive the usual mental health counseling provided through their school counselors. There is no structured curriculum for the group counseling programs but are available to all students as needed. The Lincoln Public School District also provides additional resources on specific topics such as trauma, depression and anxiety in children and adolescents, and alcohol substance use in families and provide appropriate referrals for those in need. Additionally, through organizations such as the International Council for Refugees and Immigrants (ICRI), refugee youth 7 to 18 years of age can receive educational and social support programs, after-school STEM clubs and one-on-one peer mentoring. Through the New Life Family Alliance, in addition to after-school program, boys and girls basketball program, youth are connected to youth-serving agencies that can help them effectively and successfully develop and take advantage of opportunities available to them.

INTERVENTIONS:
Behavioral: RRF4H Combination Intervention — MFG: is a family strengthening model where children and their parents sit together in groups of 8 to 10 families to discuss important issues. MFG approach provides a social support mechanism and strengthens family relationships by allowing families to share common experiences as well as effective strategies for addressing difficult issues; and focuses on reducing stigma and normalizing common experiences.
  TAHC: This is a peer-led program that allows younger students to talk with peers about important issues that they face, gain role models, and identify positive social norms from older peers. It provides age-appropriate lessons and is delivered in a structured fashion. The curriculum consists of sixteen 50-minute lessons spread out over two academic years. Topics delivered in the curriculum include substance use, positive outlook on life, forming a positive self-concept, decision making and problem solving, coping with depression, bullying and social media.
  Other Names: Virtual TeenAge Health Consultants (TAHC)
  Arms: RRF4H Combination Intervention Group

SUMMARY:
The goal of this type I hybrid effectiveness-implementation trial is to test a family strengthening (FS) model delivered through multiple family groups (MFG) combined with a virtual peer mentoring program called TeenAge Health Consultants (Virtual TAHC) aimed at addressing emotional and behavioral problems among youth born in the U.S. to parents resettled as refugees. The specific aims of the study are:

Aim 1: To systematically adapt an evidence-based family strengthening (FS) model delivered through multiple family groups (MFG) combined with a peer mentoring program (Virtual TAHC) (Goal 1).

Aim 2: To assess preliminary short- and long-term impact of the combination intervention (MFG + Virtual TAHC) on behavioral emotional disorders (aggressive behavior, antisocial behaviors, anxiety, depression, and Posttraumatic Stress Disorder [PTSD]) related to intergenerational trauma among SGRC in the trial (Goal 2).

Aim 3: Utilizing mixed methods and applying the Exploration, Preparation, Implementation, Sustainment (EPIS) framework, examine implementation strategies, facilitators, and barriers of the RRF4H intervention (Goal 3).

Participants will receive:

1. Family strengthening intervention delivered through multiple family groups (MFG) where children and one of their biological parents will participate in 16 weekly group sessions to discuss common problems and how to address them.
2. The youth in the intervention will participate in a peer mentorship program called TeenAge Health Consultants (TAHC) consisting of 16 weekly virtual sessions where they interact with other youth to learn about important topics including how to deal with conflict, stay out of trouble, deal with stress, avoid drugs and other topics.

Researchers will compare the intervention group to a control group that will receive the usual care to see if the intervention group shows improvement in symptoms compared to the usual care group.

DETAILED DESCRIPTION:
This is a type 1hybrid effectiveness-implementation trial to test a combination intervention designed to improve intergenerational trauma-related mental health symptoms among second generation refugee children (SGRC). Guided by Social Action and Family Systems theories, and applying them to the ITT framework, the proposed combination intervention consists of: family strengthening (FS) model delivered through multiple family groups (MFG) + peer mentoring program called TeenAge Health Consultants (TAHC) adapted for delivery in virtual environment (Virtual TAHC). The proposed study, titled Resettled Refugee Families for Healing (RRF4H): A Study of Intergenerational Impact of War Trauma and Resilience, will target refugee families resettled in Omaha and Lincoln, Nebraska. Using a two-arm randomized controlled trial, the investigators plan to recruit 154 children (77 per study arm), ages 14 - 17 and at least one biological parent per youth from resettled refugee communities. The intervention will be implemented over 16 weeks, with assessments at baseline, 16 weeks, and 6 months follow-up. The intervention will have the following specific aims: (1) systematically adapt an evidence-based family strengthening (FS) model delivered through multiple family groups (MFG) combined with a peer mentoring program (Virtual TAHC) (Goal 1); (2) assess preliminary short- and long-term impact of the combination intervention (MFG + Virtual TAHC) on behavioral emotional disorders (aggressive behavior, antisocial behaviors, anxiety, depression, and Posttraumatic Stress Disorder [PTSD]) related to intergenerational trauma among SGRC in the trial (Goal 2); and (3) utilizing mixed methods and applying the Exploration, Preparation, Implementation, Sustainment (EPIS) framework, examine implementation strategies, facilitators, and barriers of the RRF4H intervention (Goal 3).

ELIGIBILITY:
Inclusion Criteria for Children:

* Child born in the US
* Ages 14-17 years
* In the 9th - 12th grades
* Enrolled in one of the schools in Omaha and Lincoln, NE area Schools

Inclusion Criteria for Peer Mentors:

* Peer mentors must be students in upper class (11th or 12th grade) and
* Willing and able to serve as good role models
* Peer mentors must be nominated by community leaders

Inclusion Criteria for Parents:

* Parents must be someone resettled in the U.S. as refugee and be a biological parent of a child between the ages 14-17 years
* Parents must be ≥30 years of age

Exclusion Criteria for All Participants:

* Can understand the study procedures and/or participant rights during the informed consent process
* Unwilling or unable to commit to completing the study; 2)
* Present with emergency needs (e.g., hospitalization), needed care will be secured, rather than study participation.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 308 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in Post-Traumatic Stress Disorder (PTSD) Symptoms among adolescents | Baseline, 16 Weeks post-intervention, and 6 months
  Change in symptoms of post-traumatic stress disorder (PTSD) will be assessed using Posttraumatic Stress Disorder Reaction Index (PTSD-RI) for adolescents. PTSD scores will be dichotomized between meeting diagnostic criteria for PTSD (>=35) and not meeting diagnostic criteria for PTSD (<35).
Improvement in Post-Traumatic Stress Disorder (PTSD) Symptoms among adults | Baseline, 16 Weeks post-intervention, and 6 months
  Change in symptoms of post-traumatic stress disorder (PTSD) will be assessed using the Harvard Trauma Questionnaire (HTQ). PTSD score will be dichotomized between meeting diagnostic criteria for PTSD >=2.0 and not meeting diagnostic criteria for PTSD <2.0.
Improvement in Depression Symptoms among adults | Baseline, 16 Weeks post-intervention, and 6 months
  Changes in depression symptoms will be measured using the Hopkins symptoms checklist 25. Depression score will be dichotomized between meeting diagnostic criteria for depression (>=1.75) and not meeting diagnostic criteria for depression (<1.75).
Improvement in Depression Symptoms among adolescents | Baseline, 16 Weeks post-intervention, and 6 months
  Changes in depression symptoms will be measured using Hopkins symptoms checklist 37. There is no set clinical cut-off level, but higher score indicates symptoms severity.
Improvement in Anxiety Symptoms among adults | Baseline, 16 Weeks post-intervention, and 6 months
  Changes in anxiety symptoms will be measured using Hopkins symptoms checklist 25. Anxiety score will be dichotomized between meeting diagnostic criteria for anxiety (>=1.75) and not meeting diagnostic criteria or anxiety (<1.75)
Improvement in Anxiety Symptoms among adolescents | Baseline, 16 Weeks post-intervention, and 6 months
  Changes in depression symptoms will be measured using Hopkins symptoms checklist 37. There is no set clinical cut-off level, but higher score indicates symptoms severity.
Improvements in Antisocial Behavior Symptoms (adolescents only) | Baseline, 16 Weeks post-intervention, and 6 months
  Changes in antisocial behavior will be assessed using the Child Behavior Checklist for ages 6 to 18 years. T-scores will be dichotomized between abnormal range (T-score >=69) and normal range (T-score <69).
Improvement in Aggressive Behavior Symptoms (adolescents only) | Baseline, 16 Weeks post-intervention, and 6 months
  Changes in aggressive behavior will be assessed using the Child Behavior Checklist for ages 6 to 18 years. T-scores will be dichotomized between abnormal range (T-score >=69) and normal range (T-score <69).

SECONDARY OUTCOMES:
Improvement in Family Cohesion | Baseline, 16 Weeks post-intervention, and 6 months
  Change in family cohesion will be assessed using family cohesion scale. This is a 6-item scale with possible scores ranging from 6 to 30 and higher score indicates higher degree of family cohesion.
Improvement in Social Social Support | Baseline, 16 Weeks post-intervention, and 6 months
  Change in family and social support will be assessed using Multidimensional scale of perceived social support. Scores range from 12 to 84 with higher score indicating higher social support.
Improvement in Family and Social Support | Baseline, 16 Weeks post-intervention, and 6 months
  Change in family and social support will be assessed using University of California, Los Angeles (UCLA) Loneliness Scale, version 3. Scores range from 20 to 80 with higher score indicating higher loneliness.
Improvement in Family Communication | Baseline, 16 Weeks post-intervention, and 6 months
  Change in family communication will be assessed using Child-Adolescent Communication Scale. Two subscales: 1) degree of openness: with higher score indicating better communication (scores range from 10 to 40); and 2) extent of problems with higher score indicating more problems in parent-child communication (scores range from 10 to 50).
Improvement in Family Functioning | Baseline, 16 Weeks post-intervention, and 6 months
  Change in family functioning will be assessed using six healthy general functioning items from the McMaster Family Assessment Device with possible scores ranging from 6 to 24 and lower score indicating healthy functioning.
Mental Health Stigma | Baseline, 16 Weeks post-intervention, and 6 months
  Change in stigma symptoms will be assessed using the Paediatric Self-Stigmatization Scale. Scores range from 31 to 114 with higher score indicating high degree of stigmatization.
Improvement in Self-Concept | Baseline, 16 Weeks post-intervention, and 6 months
  Change in Self-Concept will be assessed using Tennessee Self-Concept Scale. This is a 20-item scale with scores ranging from 20 to 100 and higher score indicating higher self-concept.
Improvement in Self-efficacy | Baseline, 16 Weeks post-intervention, and 6 months
  Change in Self-Efficacy will be assessed using the General Self-Efficacy Scale, a 10-item scale with scores ranging from 10 to 40 and higher score indicating higher self-efficacy.
Improvement in Hopelessness | Baseline, 16 Weeks post-intervention, and 6 months
  Change in hopelessness will be measured using Beck Hopelessness Scale. Scores range from 20 to 40 with higher score indicating higher degree of hopelessness.
Improved peer support/relationships | Baseline, 16 Weeks post-intervention, and 6 months
  Change in peer support relationship will be assessed using Strengths and Difficulties Questionnaire (SDQ). Scores for this subscale range from 5 to 25 with higher score indicating higher degree of peer relationships.
Improved prosocial attitudes/conduct problems | Baseline, 16 Weeks post-intervention, and 6 months
  Change in prosocial attitudes/conduct problems will be measured using the Strengths and Difficulties Questionnaire (SDQ). Scores for this subscale range from 5 to 25 with higher score indicating higher degree of peer relationships.
Exposure to Potentially Traumatic Events (PTE) | Baseline, 16 Weeks post-intervention, and 6 months
  Number of traumatic events participants are exposed to will be measured using the UCLA posttraumatic stress disorder reaction index (PTSD-RI). Higher score indicates high number of traumatic events.
Exposure to Adverse Childhood Experiences (ACEs) | Baseline, 16 Weeks post-intervention, and 6 months
  Number of Adverse Childhood Experiences (ACEs) will be measured using Adverse Childhood Experience (ACEs) scale. Possible scores range from 1 to 10 with high number indicating higher ACEs score.
Change in Risk-taking Behaviors | Baseline, 16 Weeks post-intervention, and 6 months
  Change in Risk-Taking Behaviors will be assessed using the Youth Risk Behavior Survey.

OTHER OUTCOMES:
Intervention Feasibility | Baseline, 16 Weeks post-intervention, and 6 months
  Intervention feasibility will be measured using Recruitment rates; proportion eligible and enrolled (≥70% enrollment considered feasible)
Intervention Acceptability | 6 months post-intervention
  Intervention acceptability will be assessed using Client Satisfaction Questionnaire (CSQ-8; to be adapted). Scores range from 8 to 32 with higher score indicating higher degree of satisfaction/acceptability/

CONTACTS AND LOCATIONS:
Overall Officials: Nhial T Tutlam, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Nile Lutheran Church, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Once all of the data has been de-identified, cleaned, and validated, and main findings have been published, the principal investigator (PI) intends to share the data and I will ensure all mechanisms used to share data will include proper plans and safeguards for the protection of privacy, confidentiality, and security for data dissemination and reuse (e.g., all data will be thoroughly de-identified and will not be traceable to a specific study participant). Plans for archiving and long-term preservation of the data will be implemented, as appropriate.
Supporting Information: Study Protocol, Analytic Code

REFERENCES:
- [Background] Bronstein I, Montgomery P. Psychological distress in refugee children: a systematic review. Clin Child Fam Psychol Rev. 2011 Mar;14(1):44-56. doi: 10.1007/s10567-010-0081-0. PMID 21181268
- [Background] Jany L. Growing opioid use in Somali community spurs need for culturally relevant treatment. StarTribune2021
- [Background] McCleary JS, Shannon PJ, Cook TL. Connecting Refugees to Substance Use Treatment: A Qualitative Study. Soc Work Public Health. 2016;31(1):1-8. doi: 10.1080/19371918.2015.1087906. Epub 2015 Dec 14. PMID 26667046
- [Background] Gundel BE. Sudanese refugees' psychological need and mental health care: A phenomenological study of Sudanese beliefs about psychological treatment. The University of Nebraska-Lincoln; 2016
- [Background] Tutlam NT. The Impact of Maternal War Trauma on Children: A Study of South Sudanese Families Resettled in the US, Saint Louis University; 2017
- [Background] Ensor MO. South Sudanese diaspora children: Contested notions of childhood, uprootedness, and belonging among young refugees in the US. In: Contested childhoods: Growing up in migrancy. Springer, Cham; 2016:61-77.
- [Background] Kroll J, Yusuf AI, Fujiwara K. Psychoses, PTSD, and depression in Somali refugees in Minnesota. Soc Psychiatry Psychiatr Epidemiol. 2011 Jun;46(6):481-93. doi: 10.1007/s00127-010-0216-0. Epub 2010 Mar 31. PMID 20354676
- [Background] Minnesota State Epidemiological Outcomes Workgroup. Epidemiological Profile of Substance Use +Related Factors among Minnesota's Somali Youth. In: Minnesota Schools ea, ed. Saint Paul2017.
- [Background] Abur W. Settlement strategies for the South Sudanese community in Melbourne: an analysis of employment and sport participation. Melbourne: Victoria University. 2018.
- [Background] Sowey H. Are refugees at increased risk of substance misuse. Sydney: Drug and Alcohol Multicultural Education Centre. 2005
- [Background] Spencer JH, Le TN. Parent refugee status, immigration stressors, and Southeast Asian youth violence. J Immigr Minor Health. 2006 Oct;8(4):359-68. doi: 10.1007/s10903-006-9006-x. PMID 16841183
- [Background] Buchanan RL, Smokowski PR. Pathways from acculturation stress to substance use among latino adolescents. Subst Use Misuse. 2009;44(5):740-62. doi: 10.1080/10826080802544216. PMID 19308866
- [Background] Reid CA, Lorraine Beyer, Nick Crofts, Gary. Ethnic communities' vulnerability to involvement with illicit drugs. Drugs: education, prevention and policy. 2001;8(4):359-374.
- [Background] Poppitt G, Frey R. Sudanese adolescent refugees: Acculturation and acculturative stress. Journal of Psychologists and Counsellors in Schools. 2007;17(2):160-181.
- [Background] Milner K, Khawaja NG. Sudanese refugees in Australia: The impact of acculturation stress. Journal of Pacific Rim Psychology. 2010;4(1):19-29
- [Background] Fosados R, McClain A, Ritt-Olson A, Sussman S, Soto D, Baezconde-Garbanati L, Unger JB. The influence of acculturation on drug and alcohol use in a sample of adolescents. Addict Behav. 2007 Dec;32(12):2990-3004. doi: 10.1016/j.addbeh.2007.06.015. Epub 2007 Jun 9. PMID 17618064
- [Background] Priest N, Paradies Y, Trenerry B, Truong M, Karlsen S, Kelly Y. A systematic review of studies examining the relationship between reported racism and health and wellbeing for children and young people. Soc Sci Med. 2013 Oct;95:115-27. doi: 10.1016/j.socscimed.2012.11.031. Epub 2012 Dec 19. PMID 23312306
- [Background] Kellermann NP. Epigenetic transmission of Holocaust trauma: can nightmares be inherited? Isr J Psychiatry Relat Sci. 2013;50(1):33-9. PMID 24029109
- [Background] van IJzendoorn MH, Bakermans-Kranenburg MJ, Sagi-Schwartz A. Are children of Holocaust survivors less well-adapted? A meta-analytic investigation of secondary traumatization. J Trauma Stress. 2003 Oct;16(5):459-69. doi: 10.1023/A:1025706427300. PMID 14584630
- [Background] Motta R. Personal and intrafamilial effects of the Vietnam war experience. The Behavior Therapist. 1990;13:155-157.
- [Background] Roth M, Neuner F, Elbert T. Transgenerational consequences of PTSD: risk factors for the mental health of children whose mothers have been exposed to the Rwandan genocide. Int J Ment Health Syst. 2014 Apr 1;8(1):12. doi: 10.1186/1752-4458-8-12. PMID 24690436
- [Background] Bowers ME, Yehuda R. Intergenerational Transmission of Stress in Humans. Neuropsychopharmacology. 2016 Jan;41(1):232-44. doi: 10.1038/npp.2015.247. Epub 2015 Aug 17. PMID 26279078
- [Background] Isobel S, Goodyear M, Furness T, Foster K. Preventing intergenerational trauma transmission: A critical interpretive synthesis. J Clin Nurs. 2019 Apr;28(7-8):1100-1113. doi: 10.1111/jocn.14735. Epub 2019 Jan 7. PMID 30556334
- [Background] Sangalang CC, Vang C. Intergenerational Trauma in Refugee Families: A Systematic Review. J Immigr Minor Health. 2017 Jun;19(3):745-754. doi: 10.1007/s10903-016-0499-7. PMID 27659490
- [Background] Sack WH, Clarke GN, Seeley J. Posttraumatic stress disorder across two generations of Cambodian refugees. J Am Acad Child Adolesc Psychiatry. 1995 Sep;34(9):1160-6. doi: 10.1097/00004583-199509000-00013. PMID 7559310
- [Background] Daud A, Skoglund E, Rydelius PA. Children in families of torture victims: Transgenerational transmission of parents' traumatic experiences to their children. International Journal of Social Welfare. 2005;14(1):23-32.
- [Background] Caselli LT, Motta RW. The effect of PTSD and combat level on Vietnam veterans' perceptions of child behavior and marital adjustment. J Clin Psychol. 1995 Jan;51(1):4-12. doi: 10.1002/1097-4679(199501)51:13.0.co;2-e. PMID 7782473
- [Background] Dekel R, Goldblatt H. Is there intergenerational transmission of trauma? The case of combat veterans' children. Am J Orthopsychiatry. 2008 Jul;78(3):281-9. doi: 10.1037/a0013955. PMID 19123747
- [Background] Rosenheck R, Nathan P. Secondary traumatization in children of Vietnam veterans. Hosp Community Psychiatry. 1985 May;36(5):538-9. doi: 10.1176/ps.36.5.538. No abstract available. PMID 4007811
- [Background] Rosenheck R, Thomson J. "Detoxification" of Vietnam War trauma: a combined family-individual approach. Fam Process. 1986 Dec;25(4):559-70. doi: 10.1111/j.1545-5300.1986.00559.x. PMID 3817129
- [Background] Roberts AL, Galea S, Austin SB, Cerda M, Wright RJ, Rich-Edwards JW, Koenen KC. Posttraumatic stress disorder across two generations: concordance and mechanisms in a population-based sample. Biol Psychiatry. 2012 Sep 15;72(6):505-11. doi: 10.1016/j.biopsych.2012.03.020. Epub 2012 Apr 21. PMID 22521146
- [Background] Tutlam NT, Flick LH, Xian H, Matsuo H, Tutdeal N, Glowinski A. Emotional and Behavioral Disorders Among US-Born Children of South Sudanese Parents Resettled as Refugees. Global Social Welfare. 2022:1-10.
- [Background] Tutlam NT, Flick LH, Xian H, Matsuo H, Glowinski A, Tutdeal N. Trauma-Associated Psychiatric Disorders Among South Sudanese Dinka and Nuer Women Resettled in the USA. Global Social Welfare. 2020;7(3):189-199.
- [Background] Tutlam NT, Liu Y, Nelson EJ, Flick LH, Chang JJ. The Effects of Race and Ethnicity on the Risk of Large-for-Gestational-Age Newborns in Women Without Gestational Diabetes by Prepregnancy Body Mass Index Categories. Matern Child Health J. 2017 Aug;21(8):1643-1654. doi: 10.1007/s10995-016-2256-x. PMID 28092059
- [Background] Tutlam NT, Chang JJ, Byansi W, Flick LH, Ssewamala FM, Betancourt TS. War-Affected South Sudanese in Settings of Preflight, Flight, and Resettlement: a Systematic Review and Meta-analysis of Trauma-Associated Mental Disorders. Glob Soc Welf. 2024 Sep;11(3):193-210. doi: 10.1007/s40609-022-00227-w. Epub 2022 Jul 18. PMID 39588290
- [Background] Ssewamala FM, Bermudez LG, Neilands TB, Mellins CA, McKay MM, Garfinkel I, Sensoy Bahar O, Nakigozi G, Mukasa M, Stark L, Damulira C, Nattabi J, Kivumbi A. Suubi4Her: a study protocol to examine the impact and cost associated with a combination intervention to prevent HIV risk behavior and improve mental health functioning among adolescent girls in Uganda. BMC Public Health. 2018 Jun 5;18(1):693. doi: 10.1186/s12889-018-5604-5. PMID 29871619
- [Background] Chacko A, Gopalan G, Franco L, Dean-Assael K, Jackson J, Marcus S, Hoagwood K, McKay M. Multiple Family Group Service Model for Children With Disruptive Behavior Disorders: Child Outcomes at Post-Treatment. J Emot Behav Disord. 2015 Jun;23(2):67-77. doi: 10.1177/1063426614532690. PMID 26316681
- [Background] Gopalan G, Bornheimer LA, Acri MC, Winters A, O'Brien KH, Chacko A, McKay MM. Multiple family group service delivery model for children with disruptive behavior disorders: Impact on caregiver stress and depressive symptoms. J Emot Behav Disord. 2018 Sep;26(3):182-192. doi: 10.1177/1063426617717721. Epub 2017 Jul 10. PMID 30505141
- [Background] Weine S, Kulauzovic Y, Klebic A, Besic S, Mujagic A, Muzurovic J, Spahovic D, Sclove S, Pavkovic I, Feetham S, Rolland J. Evaluating a multiple-family group access intervention for refugees with PTSD. J Marital Fam Ther. 2008 Apr;34(2):149-64. doi: 10.1111/j.1752-0606.2008.00061.x. PMID 18412823
- [Background] Keiley MK, Zaremba-Morgan A, Datubo-Brown C, Pyle R, Cox M. Multiple-Family Group Intervention for Incarcerated Male Adolescents Who Sexually Offend and Their Families: Change in Maladaptive Emotion Regulation Predicts Adaptive Change in Adolescent Behaviors. J Marital Fam Ther. 2015 Jul;41(3):324-39. doi: 10.1111/jmft.12078. Epub 2014 May 8. PMID 24809985
- [Background] Clarahan W, Christenson JD. Family involvement in the treatment of adolescent substance abuse. In: Family therapy with adolescents in residential treatment. Springer; 2017:231-243
- [Background] Jackson JM. Multi-family groups for multi-stressed families: Initial outcomes and future implications. Research on Social Work Practice. 2015;25(5):537-548
- [Background] Cuijpers P. Peer-led and adult-led school drug prevention: a meta-analytic comparison. J Drug Educ. 2002;32(2):107-19. doi: 10.2190/LPN9-KBDC-HPVB-JPTM. PMID 12206061
- [Background] Matz AK. Commentary: Do youth mentoring programs work? A review of the empirical literature. Journal of juvenile justice. 2014;3(2):83.
- [Background] Tolan P, Henry D, Schoeny M, Bass A, Lovegrove P, Nichols E. Mentoring interventions to affect juvenile delinquency and associated problems: A systematic review. Campbell Systematic Reviews. 2013;9(1):1-158.
- [Background] Marsch LA, Borodovsky JT. Technology-based Interventions for Preventing and Treating Substance Use Among Youth. Child Adolesc Psychiatr Clin N Am. 2016 Oct;25(4):755-68. doi: 10.1016/j.chc.2016.06.005. Epub 2016 Aug 3. PMID 27613350
- [Background] First MB. QuickSCID-5: Quick Structured Clinical Interview for DSM-5 Disorders. American Psychiatric Association Publishing; 2021.
- [Background] Omaha Public Schools. Student and Community Services: School Counseling. 2021; https://www.ops.org/site/Default.aspx?PageID=557. Accessed October 15, 2021
- [Background] Lincoln Public Schools. Student Services: Social Workers. 2021; https://home.lps.org/socialworkers. Accessed October 15, 2021
- [Background] International Council for Refugees and Immigrants. Youth Services. 2022; https://icrius.org/programs/youth-services/. Accessed October 15, 2022.
- [Background] New Life Family Alliance. Youth Programs. 2022; https://nlfaomaha.org/youth-programs. Accessed October 15, 2022
- [Background] McKay MM, Gonzales JJ, Stone S, Ryland D, Kohner K. Multiple family therapy groups: A responsive intervention model for inner city families. Social Work with Groups. 1995;18(4):41-56
- [Background] McKay MM, Gonzales J, Quintana E, Kim L, Abdul-Adil J. Multiple family groups: An alternative for reducing disruptive behavioral difficulties of urban children. Research on Social Work Practice. 1999;9(5):593-607.
- [Background] Wilhelm AK, McRee AL, Bonilla ZE, Eisenberg ME. Mental health in Somali youth in the United States: the role of protective factors in preventing depressive symptoms, suicidality, and self-injury. Ethn Health. 2021 May;26(4):530-553. doi: 10.1080/13557858.2018.1514451. Epub 2018 Aug 24. PMID 30141350
- [Background] Betancourt TS, Berent JM, Freeman J, Frounfelker RL, Brennan RT, Abdi S, Maalim A, Abdi A, Mishra T, Gautam B, Creswell JW, Beardslee WR. Family-Based Mental Health Promotion for Somali Bantu and Bhutanese Refugees: Feasibility and Acceptability Trial. J Adolesc Health. 2020 Mar;66(3):336-344. doi: 10.1016/j.jadohealth.2019.08.023. Epub 2019 Nov 5. PMID 31699604
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Diggle P, Heagerty P, Liang K, Zeger S. Analysis of Longitudinal Data: Oxford University Press.[Google Scholar]. 2002
- [Background] Management Information System for Individual Development Accounts: A Feasibility Study (CSD Report No. 01-21) [computer program]. St. Louis, MO: Washington University, Center for Social Development; 2001
- [Background] MIS IDA Operations Manual: Management Information System for Individual Development Accounts, Version 5 [Computer Software Manual] [computer program]. St. Louis, MO: Washington University, Center for Social Development; 2006
- [Background] Luellen JK, Shadish WR, Clark MH. Propensity scores: an introduction and experimental test. Eval Rev. 2005 Dec;29(6):530-58. doi: 10.1177/0193841X05275596. PMID 16244051
- [Background] van der Laan M, Rose S. Targeted Learning: Causal Inference for Observational and Experimental Data. New York, NY: Springer; 2011.
- [Background] Enders CK. Applied Missing Data Analysis. New York: Guilford Press; 2010.
- [Background] Little RJA, Rubin DB. Statistical Analysis with Missing Data. New York: John Wiley and Sons; 2002.
- [Background] Collins LM, Schafer JL, Kam CM. A comparison of inclusive and restrictive strategies in modern missing data procedures. Psychol Methods. 2001 Dec;6(4):330-51. PMID 11778676
- [Background] Cro S, Morris TP, Kenward MG, Carpenter JR. Sensitivity analysis for clinical trials with missing continuous outcome data using controlled multiple imputation: A practical guide. Stat Med. 2020 Sep 20;39(21):2815-2842. doi: 10.1002/sim.8569. Epub 2020 May 17. PMID 32419182
- [Background] SAS Institute. BASE SAS 9.4 Procedures Guide. Cary, NC: SAS Institute, Inc.; 2013.
- [Background] Westfall PH, Young SS. Resmpling Based Multiple Testing: Examples and Methods for p-value Adjustment. New York, NY: John Wiley and Sons; 1993
- [Background] Rodriguez G, Goldman N. An Assessment of Estimation Procedures for Multilevel Models with Binary Responses. Journal of the Royal Statistical Society Series a-Statistics in Society. 1995;158:73-89.
- [Background] Haybittle JL. Repeated assessment of results in clinical trials of cancer treatment. Br J Radiol. 1971 Oct;44(526):793-7. doi: 10.1259/0007-1285-44-526-793. No abstract available. PMID 4940475
- [Background] Peto R, Pike MC, Armitage P, Breslow NE, Cox DR, Howard SV, Mantel N, McPherson K, Peto J, Smith PG. Design and analysis of randomized clinical trials requiring prolonged observation of each patient. II. analysis and examples. Br J Cancer. 1977 Jan;35(1):1-39. doi: 10.1038/bjc.1977.1. PMID 831755
- [Derived] Tutlam NT, Liyew TW, Betancourt TS, Powell BJ, Guo S, McKay M, Ssewamala FM. Type I hybrid effectiveness-implementation randomised controlled trial to address intergenerational impact of war trauma and resilience among second-generation refugee children in the USA: Resettled Refugee Families for Healing (RRF4H) study protocol. BMJ Open. 2025 Oct 16;15(10):e108824. doi: 10.1136/bmjopen-2025-108824. PMID 41101964